CLINICAL TRIAL: NCT00425867
Title: PAR Family Polymorphisms and Placental Invasion Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Other Study IDs: PAR1 polymorphisms
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Miscarriage, Recurrent; Premature Labor
Keywords: PAR1 gene; polymorphisms; abortions; reccurent abortions; premature delivery
MeSH Terms: conditions — Abortion, Habitual; Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

INTERVENTIONS:
Behavioral: PAR1 polymoprhisms and placental invasion

SUMMARY:
The present study will be undertaken to establish whether genetic variations of PAR1 could be involved in the occurrence of any of the "placental syndromes" of preterm delivery, preeclampsia, and/or small for gestational age babies and recurrent pregnancy loss.

DETAILED DESCRIPTION:
Polymorphisms of Protease Activated Receptor 1 and adverse pregnancy outcomes Protease Activated Receptor 1 (PAR1), the main thrombin receptor on vascular cells (Coughlin,1999), plays a critical role in orchestrating human placentation based on temporally and spatially constrained PAR1 expression in the normal invasive trophoblasts (O'Brien et al, 2003) and its overexpression in pathological invasive trophoblast (Even-Ram et al, 2003).

Various proteases of the PAR family as well as matrix metalloproteinases have been implicated in ancillary regulation of cancer metastases and tumor-related angiogenesis. PAR1 in particular has been proposed to be involved in invasive processes of various cancers (Ruf & Mueller, 2006; Boire et al, 2005). Similarly, it might be surmised that remodeling of the placenta microenvironment as well as the requisites of trophoblast invasiveness may be PAR1 sensitive (Grisaru-Granovsky et al, 2005). Therefore, one might hypothesize that PAR1 gene variability may be involved in early placentation and that adverse pregnancy outcomes of the "placental syndromes" may have their origin in PAR1 dysregulation.

Study Design: This is a prospective case-control pilot study. Subject enrolment and data collection will be performed via the Admission Service of the Division for Maternal & Fetal Medicine in a large tertiary obstetrics department in Jerusalem, Israel. Demographic data including maternal characteristics, past reproductive history, and information about previous complications during pregnancy, delivery and the neonatal period will be culled. The blood samples will be collected at routine admission after obtaining informed consent by the physician on the floor.

Four groups are described: patients with spontaneous preterm delivery of a singleton before 35 weeks of gestation; patients with a singleton pregnancy complicated by preeclampsia diagnosed according the Working Group Criteria (2000); patients who deliver a small for gestational age (SGA) singleton defined as a birth weight below the 10th percentile for the gestational age according to the Israeli growth curves (Dollberg et al, 2005); and for comparison, patients who deliver a singleton at term with appropriate size for gestational age. Patients who suffer delivery with intrauterine fetal demise and/or neonates with malformations will be excluded.

Maternal and umbilical cord blood samples (in 0.11mol/l sodium tri citrate) will be paired. DNA will be prepared from white blood cells by standard techniques and subsequently stored at -4°C for batched analysis. The laboratory staff will be blinded as to the clinical status of the samples.

Polymorphism analysis will be performed for the following polymorphisms of the PAR1 gene: [-1426CT], [506 insertion of 13 bp],[IVS-14A/T]: as per standard PCR techniques using appropriate restriction endonucleases (Arnaud et l, 2000).

ELIGIBILITY:
Inclusion Criteria:

* Women with reccurent abortions unexplained
* Premature delicery

Exclusion Criteria:

* Term pregnancies
* Abortion that the cause is known

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2007-03; Study Completion 2007-11

CONTACTS AND LOCATIONS:
Overall Officials: Sorina Grisaru, MD, Principal Investigator — Shaare Zedek Medical Center

REFERENCES:
- See also: Related Info — http://ncbi.nlm.nih.gov
- See also: Related Info — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?db=pubmed&cmd=Retrieve&dopt=AbstractPlus&list_uids=17100658&query_hl=5&itool=pubmed_docsum
- See also: Related Info — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?db=pubmed&cmd=Retrieve&dopt=AbstractPlus&list_uids=17097558&query_hl=5&itool=pubmed_docsum
- See also: Related Info — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?db=pubmed&cmd=Retrieve&dopt=AbstractPlus&list_uids=16710477&query_hl=15&itool=pubmed_docsum
- See also: Related Info — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?db=pubmed&cmd=Retrieve&dopt=AbstractPlus&list_uids=16081834&query_hl=15&itool=pubmed_docsum